CLINICAL TRIAL: NCT05363449
Title: An Open Label, Parallel Group Comparison Study To Evaluate the Safety Tolerability, and Pharmacokinetics of UHE-103 Cream Versus Naftin Cream in Subjects With Tinea Cruris and/or Tinea Pedis Under Maximal Use Conditions
Brief Title: Safety, Tolerability, and Pharmacokinetics of UHE-103 Cream in Subjects With Tinea Cruris and/or Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 146-9252-102
Record Dates: First submitted 2022-03-10; First posted 2022-05-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Tinea Cruris; Tinea Pedis
MeSH Terms: conditions — Tinea Cruris; Tinea Pedis | interventions — naftifine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UHE-103 Cream (Experimental): Subjects will apply at least a total of 4 grams* of the test article, covering both feet twice daily for 2 weeks
  Interventions: Drug: UHE-103 Cream
- Naftin (naftifine hydrochloride) Cream, 2% (Active Comparator): Subjects will apply at least a total of 5 grams* of the test article, covering the interdigital areas of both feet and to the groin once daily for 2 weeks
  Interventions: Drug: Naftin (naftifine hydrochloride) Cream

INTERVENTIONS:
Drug: UHE-103 Cream — UHE-103 is an investigational combinational therapy containing keratolytic and antifungal
  Arms: UHE-103 Cream
Drug: Naftin (naftifine hydrochloride) Cream — Naftin (naftifine hydrochloride) Cream, 2%. Topical cream containing active drug
  Arms: Naftin (naftifine hydrochloride) Cream, 2%

SUMMARY:
This Phase 1 study has been designed to determine the safety, tolerability and pharmacokinetics (PK) of UHE 103 Cream compared to Naftin Cream, 2% under maximal use conditions for 2 weeks treatment in subjects with tinea cruris and/or tinea pedis

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female 18 years of age or older.
2. Subject has provided written informed consent.
3. Subject has a clinical diagnosis of moccasin-type tinea pedis with at least moderate scaling on at least 1 foot at Visit 1/Screening;
4. Subject has a clinical diagnosis of interdigital tinea pedis with at least moderate scaling on at least 1 foot (without moccasin-type tinea pedis) and tinea cruris at Visit 1/Screening.
5. Subject is willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has any skin pathology or condition that could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
3. Subject has any clinically significant medical abnormality or history of chronic disease (cardiovascular, gastrointestinal, neurological, hematopoietic, immunosuppression [HIV], hepatic [Hepatitis B or C], psychological, renal systems, or respiratory), including conditions (e.g., gastrointestinal surgery) that may interfere with the absorption, metabolism, or excretion of investigational product.
4. Subject has used any of the following topical products on the feet or groin within 4 weeks of Visit 2/Enrollment: antifungals, antibacterials, or corticosteroid therapy.
5. Subject has applied any topical naftifine products to any part of their body within 4 weeks of Visit 2/Enrollment.
6. Subject has used topical keratolytics (e.g., urea, ammonium lactate, salicylic acid) on the feet or groin within 1 week of Visit 2/Enrollment.
7. Subject has used any other topical products on the feet or groin within 24 hours of Visit 2/Enrollment including, but not limited to non-medicated moisturizers, antipruritics, analgesics, anesthetics, etc.
8. Subject has received systemic antifungal therapy within 8 weeks or 5 half lives of the antifungal (whichever is longer) of Visit 2/Enrollment.
9. Subject is currently enrolled in an investigational drug, biologic, or device study.
10. Subject has previously been enrolled in a study for UHE-103.
11. Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to Visit 2/Enrollment.
12. Subject has a history of sensitivity to any of the ingredients in the test articles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Baseline up to Day 16
  Percentage of subjects with any local and systemic AEs defined as "possibly" or "probably" or "definitely" related by the investigator.
Local Skin Reactions (LSRs) | Day 16
  Percentage of subjects with presence of any of the following LSRs at the end of the study: burning/stinging, edema, and oozing/vesiculation/crusting.
AUC (0-12 hours) | Day 15
  Defined as the area concentration-time curve (AUC) of the active antifungal drug from time 0 to 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics Inc. (CRO)
Locations (5):
- United States (5):
  - Site #1, San Diego, California
  - Site #5, Thousand Oaks, California
  - Site #2, Austin, Texas
  - Site #3, College Station, Texas
  - Site #4, Houston, Texas

IPD SHARING:
Plan to Share IPD: No